CLINICAL TRIAL: NCT03256500
Title: Transcranial Direct Current Stimulation for the Treatment of Delirium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: North Florida/South Georgia Veterans Health System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB201400807
Record Dates: First submitted 2017-07-24; First posted 2017-08-22 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Delirium; Confusion
MeSH Terms: conditions — Delirium; Confusion | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- tDCS administered (Experimental): Subjects will receive stimulation via tDCS (Transcranial Direct Current Stimulation) for 20 minutes per day, 5 days per week, for 1 week.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham tDCS administered (Sham Comparator): Subjects will receive sham tDCS (Transcranial Direct Current Stimulation) for 20 minutes per day, 5 days per week, for 1 week.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — One half of the subjects will receive sham and the other half will receive tDCS. The Soterix Medical 1x1 line of low-intensity tDCS stimulators which we plan to use is designed to generate low levels of direct current current between one anode and one cathode placed on the body. The current enters the body through the positive electrode, the anode exits the body through the negative electrode, the cathode. The accessories provided with the device allow for simple and comfortable positioning of the electrodes on the body.
  Other Names: tDCS

SUMMARY:
Delirium is induced by changes in cortical excitability and transcranial direct current stimulation (tDCS), by using weak electrical fields, can modulate cortical excitability and spontaneous firing activities in the stimulated region by shifting the resting membrane. One half of the subjects will receive stimulation via tDCS and the other half will receive sham tDCS for 20 minutes per day, 5 days per week, for 1 week. Symptoms will be monitored using the Confusion Assessment Method.

DETAILED DESCRIPTION:
Hospitalized patients with delirium, who are over age 21, will be the subjects for this research study. This will include both men and women at the Malcom Randall Veterans Affairs Hospital. The presence of delirium will be determined by the "Confusion Assessment Method (CAM)" which is a standardized evidence-based tool that enables clinicians to identify patients who are suffering with delirium. The CAM and the CAM-ICU have been reported to have a sensitivity of 94-100% with a specificity of 89-95%, together with a high inter-rater reliability (Wei, Fearing, Eliezer, Sternberg, & Inouye, 2008).

Patients with agitation at the moment of the procedure, pregnancy or patients with history of epilepsy or show evidence of epilepsy on their EEG will be excluded.

As part of their routine medical care all participants will be fully evaluated for the possible causes of delirium including: neurological disorders (CT or MRI, EEG, possible LP); failure of vital organs (cardiac, hepatic, renal, pulmonary), metabolic disorders (e.g. abnormalities of blood chemistries), endocrine disorders (e.g., abnormal thyroid function tests), infections (e.g., urinary, pulmonary, sepsis), toxins-drugs-medications, and deficiency states (B1, B12, etc). These conditions will be treated accordingly by their primary provider. There will be no change in the rest of the care that the patient will get when they get hospitalized.

Because patients with delirium lack the capacity to consent, the consent will be obtained from a legally authorized representative who is usually the spouse, adult child, a relative or a close friend. The legally authorized representative or guardian advocate who can make decisions on the patient's behalf, will be appointed by the legal authorities. They can be a health care surrogate/agent appointed by the person in a Durable Power of Attorney for Health Care (DPAHC) or similar document. The legally authorized representative can also be a court appointed guardian. If the patient/patient's legal representative decides to participate in the study, the Principal Investigator will collect private information about the patient's health, which is called Protected Health Information (PHI). The protected health information will be then be coded and each subject will be given a unique identification number before entering it into the password protected folder on the server. Once eligibility is determined, the information is obtained from the medical records regarding psychiatric disorders, neurological conditions, cardiac conditions, current medications, study results, age < 89 in numerical values, sex, education level and details regarding any tests or procedures done.

A neurocognitive assessment will be done on all the patients identified as potential subjects for the study. The assessment will be done by Uma Suryadevara, Colleen Campbell, Ronald Shorr, Kenneth Heilman, Laurence Solberg, Andrew Pierce or Joseph Thornton. After the assessment is done, subjects are assigned into two groups, one group that gets the sham and group that gets the real treatment. One half of the subjects will receive sham and the other half will receive tDCS. The Soterix Medical 1x1 line of low-intensity tDCS stimulators which we plan to use is designed to generate low levels of direct current between one anode and one cathode placed on the body. The current enters the body through the positive electrode, the anode exits the body through the negative electrode, the cathode. The accessories provided with the device allow for simple and comfortable positioning of the electrodes on the body. The procedure will be done by Uma Suryadevara who went through the training and is certified and Colleen Campbell will activate the sham in some patients. Laurence Solberg, Ronald shorr, Andrew Pierce and Joseph Thornton will do the procedure after being trained. Adam Woods is the expert in tDCS and has been teaching this procedure for sometime now and will help us with the process. The transcranial Direct Current Stimulator has the option of activating or deactivating the 'sham'. All participants will be treated with sham or real tDCS for 20 minutes per day, 5 days per week, for 1 week during their hospitalization. The person performing the neurocognitive assessment will be unaware if the participant is receiving sham or tDCS. The electrodes will be placed over the left and right frontal lobes, near the dorsolateral prefrontal cortex, (anode on the left and cathode on the right) using the International 10-20 system as a guide for electrode placement. (Poreisz et al., 2007; Nitsche et al, 2012. tDCS utilizes either two saline-soaked sponge or electrode gel coated electrodes affixed to the scalp, which causes a weak electrical current. The maximum output of the current is 2 milliamp and each electrode has an area of 25-35 cm^2. For stimulation in the experimental condition, a current of 1.0-2.0 milliamps will be used, which is gradually increased and decreased to achieve this target current over 30 seconds. Vitals will be taken before and after tDCS treatments. Both before stimulation and after stimulation on each day, as well as daily one week after stimulation, subjects will undergo an assessment for change in symptoms using the Memorial Delirium Assessment Scale (MDAS). Since the effects of the stimulation may last for a short time post stimulation testing will begin approximately 5 minutes after the stimulation and be completed within one hour. Testing will also be done one more time later that afternoon to measure the change in symptoms.

The coded information and the details of the treatment will be stored on a computer server with secure passwords. This information will then be used to test the effects of transcranial Direct Current Stimulation on the symptomatic treatment of delirium. The neurocognitive tests which include both the Confusion Assessment Method and the Memorial Delirium Assessment Scale will be used to assess the symptomatic improvement. Once this information is collected, it will be a part of the research record for the study. This information will be retained according to the VA policies. The subjects will get the rest of the treatment as usual. For example, any infections will be treated, electrolyte abnormalities will be corrected, offending agents like drugs or toxins will be discontinued, deficiencies will be corrected. If there is any failure of vital organs or if there are any neurological disorders, appropriate treatments will be provided as per standards. The patients will then be discharged as appropriate.

Procedures for recruiting and consenting:

Target population: Hospitalized patients with an established diagnosis of delirium using the 'Confusion Assessment Method'.

Delirium is commonly associated with increased mortality and morbidity. It is also associated with prolonged hospitalization, increased nursing demands and need for use of physical and pharmacological restraints. Patients with delirium represent a vulnerable population for who we don't have many successful treatment options. Hence, any successful symptomatic treatment that would decrease the severity will be valuable.

Patients who are admitted to the inpatient unit, with a diagnosis of delirium based on the 'Confusion Assessment Method', are identified by the treating physician. Once the guardian advocate or legally authorized representative is appointed by the legal authorities, consent will be obtained for their participation in research by the physician. The guardian advocate or legally authorized representative is usually the spouse, adult child, a relative or a close friend. They will be given all information about the study, who to call for questions, why the study is being done, what to expect if they participate in the study and how long the study will last. They will also be given the risks and benefits of this study, possible adverse reactions, the information that will be collected and who will have access to it. They will also be made aware of the option of withdrawing from the study at any point. Once they withdraw the health information will not be collected.

If the patient/patient's legal representative decides to participate in the study, the Principal Investigator will collect private information about the patient's health, which is called PHI. (Protected Health Information). The protected health information will be then be coded before entering it into the password protected folder on the server. The information will be collected and shared with others involved in the research to determine eligibility. The information is obtained from the medical records regarding psychiatric disorders, neurological conditions, cardiac conditions, current medications, study results, age < 89 in numerical values, sex, education level and details regarding any tests or procedures done.

The information will be stored on a computer server with secure passwords. This information will then be used to test the effects of transcranial Direct Current Stimulation on the symptomatic treatment of delirium. The neurocognitive tests which include both the Confusion Assessment Method and the Memorial Delirium Assessment Scale will be used to assess the symptomatic improvement. Once this information is collected, it will be a part of the research record for the study. People who will have access to this information will be the Principal Investigator and research staff associated with the project.

While obtaining the informed consent, it will be explained to the legal authorized representative that they are not required to sign the consent and the refusal will not affect the standard treatment in any way. During the hospitalization, the participants and the non-participants will continue to get the standard treatment for delirium. The providers will evaluate for the cause of the delirium by: getting blood chemistries to rule out metabolic disorders, ruling out infections (e.g., urinary, pulmonary, sepsis), toxins-drugs-medications, deficiency states like B1, B2 etc, failure of vital organs (cardiac, hepatic, renal, pulmonary), neurological disorders using a CT or MRI, EEG, Lumbar Puncture if indicated. If any treatable cause is identified, it will be managed accordingly. Meanwhile the patient will be assessed for nutritional status, reorientation techniques will be used, sensory deficits will be corrected if present. One of the hypothesis for the pathophysiology of delirium is changes in cortical excitability; this research intervention can modulate cortical excitability and spontaneous firing activities in the stimulated region by shifting the resting membrane potential leading to symptomatic improvement in a patient with delirium.

Because Delirium is a condition that causes fluctuation in cognition, it can also cause fluctuating decision making capacity. The psychiatrists will evaluate for decision making capacity on an ongoing basis during the study. If it any point, the subject regains the capacity to consent, we will go over the consenting process again with the subject. At that point if the subject decides to withdraw from the study, the decision will be respected and if not, the study will continue as before.

The neurocognitive assessments will be done prior to and after the treatments if they decide to participate.

Statistical Analysis:

The major dependent variable will be the score on the CAM and the MDAS (modeled as a continuous variable). We will perform a mixed models analysis which will compare the trajectory of CAM and MDAS score among Experimental Participants versus Control Participants. Because this is a pilot/exploratory study, no sample size calculations are included in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with presence of delirium, confirmed by "Confusion Assessment Method". Age > 21 years old Hospitalized at the Malcom Randall Veterans Affairs Hospital. Number of patients who will be recruited: 100

Exclusion Criteria:

* Patients with agitation. Pregnancy Patents with a history of epilepsy or have evidence of epilepsy on their EEG. Implanted devices anywhere in the body Unstable medical conditions like uncontrolled Diabetes, Hypertension Unconscious patients

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-12-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in signs and symptoms of delirium | Time points at which the measurement will be done is within 5 minutes to an hour after procedure and another one will be done 4 to 5 hours later.
  Negative screens for delirium for at least 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Uma Suryadevara, MD, Principal Investigator — Malcom Randall VAMC
Locations (1):
- Malcolm Randall Veterans Affairs Medical Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.